CLINICAL TRIAL: NCT05018377
Title: Effectiveness and Safety of Percutaneous Adhesiolysis Using Rac'z Catheter Versus Navi Catheter in Management of Failed Back Surgery Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Saeid Metwaly Abouelyazid Elsawy, lecturer of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: saeid
Record Dates: First submitted 2021-03-15; First posted 2021-08-24 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Raj'z catheter (Active Comparator)
  Interventions: Procedure: Racz adhesolysis
- NAVI catheter (Active Comparator)
  Interventions: Device: NAVI adhesolysis

INTERVENTIONS:
Procedure: Racz adhesolysis — adhesiolysis in failed back surgery
  Arms: Raj'z catheter
Device: NAVI adhesolysis — adhesiolysis in failed back surgery
  Arms: NAVI catheter

SUMMARY:
In the past decade, spine surgery rates have dramatically increased in parallel to those of other procedural interventions. Persistent pain is a common occurrence after spine surgery, with the most commonly quoted prevalence rates ranging from 10% to 40%. This pain can be classified into failure to alleviate baseline pain, pain resulting from complications (e.g., arachnoiditis and epidural adhesions), and pain that ensues several years later as a sequele to alterations in spinal architecture and biomechanics (e.g., adjacent segment discogenic or facetogenic pain) which is called failed back surgery syndrome ( FBSS )

DETAILED DESCRIPTION:
By observing adhesions directly, the lysis of scar tissue can be carried out mechanically using some percutaneous techniques as insertion of catheters as Rac'z catheter (thin in calibre) which will be inserted through the skin under fluoroscopy guidance or using NAVI catheter (large in calibre) either fluoroscopy guided or using thin epiduroscopy. Adhesions can be disintegrated and their evaluation scores may improve.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of lumbar surgery of at least 6 months duration in the past.
* Patients over the 18 years of age.
* History of persistent function-limiting lower extremity pain aggravated by "dural tug" (observed when the patient, sitting on the exam table with legs stretched out, bends forward, bringing on the back pain) with or without low back pain of at least 6 months duration after failure of conventional conservative management in most patients including NSAIDS, muscle relaxants (tizanidine, magnesium sulphate) and pregabalin.
* Patients who are competent to understand the study protocol and provide voluntary, written informed consent and participate in outcome measurements.

Exclusion Criteria:

* Unstable or heavy opioid use.
* Uncontrolled psychiatric disorders.
* Uncontrolled medical illness.
* Any conditions that could interfere with the interpretation of the outcome assessments.
* Pregnant or lactating women.
* Patients with a history or potential for adverse reaction(s) to local anaesthetics or steroid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-08-13 (Actual)

PRIMARY OUTCOMES:
numerical rating scale | 12 months
  The VAS score was used that has 0-10 points. The 0 point represents the painless state and a score from 1 to 3 points represents mild pain, from 4 to 6 points represents moderate pain and from 7 to 10 points represents severe pain.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | 12 month
  0 - 100% disability; minimal disability = 0% to either bed-bound or exaggerating symptoms = 100%)
pregabalin consumption | 12 month
  amount of pregabalin consumed by the patient per day

CONTACTS AND LOCATIONS:
Locations (1):
- Saeid Metwaly Elsawy, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
may i share it